CLINICAL TRIAL: NCT01287299
Title: Dietary Glycemic Load & Metabolism in Obese Pregnant Women
Brief Title: Glycemic Load, Metabolism & Obesity in Pregnancy
Acronym: PANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: University of California, San Francisco (Other); University of California, Davis (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2500-080; R01HD046741 (NIH)
Record Dates: First submitted 2011-01-30; First posted 2011-02-01 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Insulin Resistance
Keywords: pregnancy; obesity; diet glycemic load; body composition; body fat; gestational weight gain; insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance; Gestational Weight Gain | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Glycemic Load Diet (Experimental): Counseled to consume a diet with a low or higher intake of carbohydrate sources that cause rapid or significant intakes in blood glucose. The average glycemic load of the diet should be less than 55 per 1000 calories or greater than 55 per 1000 calories.
  Interventions: Other: Low Glycemic Load diet
- Low Fat Diet (Experimental): Pregnant women were counseled to consume a diet providing less that 25% of the energy as fat.
  Interventions: Other: Low Fat Diet

INTERVENTIONS:
Other: Low Glycemic Load diet — Pregnant women were counseled to consume a diet with a glycemic load per 1000 kcal of less than 55.
  Other Names: LGL Diet
  Arms: Low Glycemic Load Diet
Other: Low Fat Diet — Pregnant women were counseled to consume diets providing less than 25% of the energy as fat.
  Other Names: LF Diet
  Arms: Low Fat Diet

SUMMARY:
The purpose of the study is to determine if a low glycemic load diet reduces the gain of body fat and insulin resistance during the last half of pregnancy in obese women.

DETAILED DESCRIPTION:
Obese women will be recruited to participate in the study between 14-18 weeks gestation. After determining usual dietary intakes, visceral fat thickness, and the metabolic response to a 100g oral glucose tolerance test (OGTT) at 20 weeks gestation, 45 of the women will be randomly assigned to a low glycemic load (GL) diet and 65 women to a regular low fat diet (current standard care). They will follow their assigned diet for the last 20 weeks of gestation. A dietitian will advise the women and will monitor them throughout the study. At 28 and 34 weeks gestation, the women will come to the General Clinical Research Center (GCRC) at San Francisco General Hospital in the fasting state and the hormonal and metabolic response will be measured to another 100g oral glucose tolerance test (OGTT), and total body fat will be measured. Additional measurements include: 1) longitudinal measurements of maternal visceral fat thickness and fetal size and adiposity at 20 and 34 weeks gestation by ultrasound, 2) collection of cord blood and placental tissue, and 3) measurement of neonatal body composition by dual-energy x-ray absorptiometry and anthropometry at 2-3 weeks of age. Birth outcome data for mother and infant will be collected. To determine the metabolic response to the study diet, 25 women from each of the two diet groups will be assigned to a metabolic subsample for measuring rates of hepatic glucose production and lipolysis at 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

* >35% body fat
* 18 to 40 years of age
* speak English or Spanish

Exclusion Criteria:

* have diabetes prior to pregnancy
* diagnosed with GDM in current pregnancy
* smoke
* abuse alcohol or drugs
* have a metabolic disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
maternal body fat gain | 20-34 weeks gestation
  Changes in total body fat as measured by air displacement between 20 to 34 weeks gestation

SECONDARY OUTCOMES:
Insulin Resistance | 20-34 weeks gestation
  Changes in insulin resistance measured during an oral glucose tolerance test between 20 to 34 weeks gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Janet C King, Ph.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States